CLINICAL TRIAL: NCT00273689
Title: "Pretreatment With Albuterol vs. Montelukast in Exercise Induced Bronchospasm in Children."
Brief Title: Exercise Induced Bronchospasm in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Hengameh Raisyy, Pharm.D., University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACCP
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Exercise Induced Bronchospasm
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Albuterol; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Other): This is a crossover trial- Patients get randomly assign to albuterol or singulair and then cross overed to the alternate active medication.
  Interventions: Drug: montelukast vs pretreatment with albuterol; Drug: montelukast

INTERVENTIONS:
Drug: montelukast vs pretreatment with albuterol — montelukast 5 or 10 mg once daily for 3 days vs albuterol 2 puffs, 15 minutes before exercise
  Other Names: Singulair is the brand name for montelukast.
Drug: montelukast — Montelukast 5 or 10 mg once daily for 3 days vs Albuterol inhlare 2 puffs, 15 minutes before exercise
  Other Names: Brand name for montelukast: Singulair

SUMMARY:
The purpose of the study is to test how well 2 different medications stop asthma symptoms caused by exercising. The two medications that will be tested are "pretreatment with albuterol" and montelukast (Singulair®). Although both medications are used for treating asthma, we don't know which medicine is better at stopping asthma symptoms caused by exercising.

DETAILED DESCRIPTION:
TThis is a randomized, crossover, placebo controlled trial of 30 patients, 7-17 years old with confirmed EIB. Patients will be randomized to montelukast treatment for at least 3 days or pretreatment with albuterol before an exercise challenge. Villiran and colleagues have shown that the protective effect of montelukast in treating EIB is apparent at day 3 of treatment and comparable to treatment for 4 and 8 weeks.

It is our hypothesis that pretreatment with albuterol will provide superior protection against breakthrough EIB in children with mild asthma compared to montelukast as maintenance therapy added to the current asthma regimen. Secondary aims of this study are to measure the effect of montelukast on leukotriene B4 (LTB4) concentrations as measured in EBC, and on inflammation measured by FeNO level. We hypothesize that since montelukast is a cysteinyl leukotriene receptor antagonist, patients with elevated concentration of LTB4 may have a greater response to this medication. Lastly, patients with elevated FeNO, a measure of airway inflammation respond differently to albuterol than montelukast his study is a randomized, double-blind, double-dummy, crossover clinical trial which will consist of 4 study visits and last up to 3 weeks.

Thirty children 7-17 years of age with asthma and EIB, regardless of current asthma therapy will be eligible for this trial. Patients will receive 3-7 days of therapy with either montelukast (5mg or 10 mg capsule) or placebo tablets. After 3-7 days of therapy the patients will be crossed over to receive the alternative therapy. Exercise challenges will be completed at screening, baseline, visit 3 and visit 4. All patients will have an albuterol metered-dose inhaler (MDI) to be used on an as needed basis for asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children 7-17 years of age
* Physician diagnosed asthma for at least 6 months
* EIB diagnosed by a positive exercise challenge at screening and baseline visits
* Forced expiratory volume in 1 second (FEV1) ≥ 70% of predicted at screening and baseline visit

Exclusion Criteria:

* History of cardiac dysfunction
* Unable to perform exercise challenge
* Use of montelukast

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the comparison of the effect of inhaled albuterol and oral montelukast on EIB as percent attenuation in FEV1 after exercise challenge. | Fall in FEV1 immediately after exercise

SECONDARY OUTCOMES:
Additional objectives will be to compare the differences in response to montelukast with regard to LTB4 concentrations from EBC and FeNO level | immediately after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Hengameh H Raissy, PharmD, Principal Investigator — University of New Mexico; William Kelly, PharmD, Study Director — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States